CLINICAL TRIAL: NCT06066645
Title: Multicenter, Randomized, Double-masked Trial to Evaluate the Safety and Efficacy of iDose® TR (Travoprost Intraocular Implant) in Conjunction With the Placement of iStent Infinite vs. iStent Infinite Alone in Subjects With Open-angle Glaucoma or Ocular Hypertension
Brief Title: Travoprost Intraocular Implant + iStent Infinite vs. iStent Infinite Alone
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Glaukos Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GLK-101-01
Record Dates: First submitted 2023-09-27; First posted 2023-10-04 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Glaucoma, Open-Angle
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (3):
- iDose TR (Experimental): Travoprost Intraocular Implant in subjects who had successful iStent infinite placement
  Interventions: Drug: Travoprost Intraocular Implant; Device: iStent infinite
- sham procedure (Sham Comparator): Sham surgical procedure
  Interventions: Other: Sham procedure 1; Device: iStent infinite
- iDose TR alone (Experimental): Travoprost Intraocular Implant
  Interventions: Drug: Travoprost Intraocular Implant; Other: Sham procedure 2

INTERVENTIONS:
Drug: Travoprost Intraocular Implant — anchored intracameral implant containing travoprost in subjects who successfully received iStent infinite
  Other Names: iDose TR
  Arms: iDose TR; iDose TR alone
Other: Sham procedure 1 — Sham procedure (to mimic placement of travoprost intraocular implant) in subjects who successfully received iStent infinite
  Arms: sham procedure
Device: iStent infinite — Successful iStent infinite surgery
  Arms: iDose TR; sham procedure
Other: Sham procedure 2 — Sham procedure (to mimic placement of an iStent infinite)
  Arms: iDose TR alone

SUMMARY:
Adult subjects with elevated intraocular pressure who have successfully undergone placement of iStent infinite trabecular bypass system will be randomized to receive a travoprost intraocular implant or receive a sham procedure and be followed for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of open-angle glaucoma or ocular hypertension
* qualifying IOP in the study eye

Exclusion Criteria:

* unmedicated (washed out) IOP of >36 mmHg in the study eye
* hypersensitivity to travoprost or any other components of the travoprost intraocular implant
* vertical cup/disc ratio > 0.8 in the study eye
* best spectacle corrected visual acuity of worse than 20/80 in either eye eye
* any ocular disease or condition that, in the opinion of the investigator, may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2023-09-14 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
change from baseline in mean diurnal intraocular pressure (IOP) | 3 months
  mean diurnal IOP at the 3 month visit minus mean diurnal IOP at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Glaukos Corporation
Locations (1):
- Glaukos Clinical Study Site, Colorado Springs, Colorado, United States

IPD SHARING:
Plan to Share IPD: No